CLINICAL TRIAL: NCT03082391
Title: Long-term Results of Heavy Weight Versus Medium Weight Mesh in Ventral Hernia Repair
Brief Title: Heavy Weight Versus Medium Weight Mesh in Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Rosen, Director, Comprehensive Hernia Center, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-1643
Record Dates: First submitted 2017-03-12; First posted 2017-03-17 (Actual); Results first posted 2022-06-22 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Ventral Hernia
Keywords: Ventral Hernia Repair; Heavy weight Mesh; Medium weight Mesh
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Heavy weight Mesh (Active Comparator): Intervention: Patients will undergo ventral hernia repair with implantation of a heavy weight mesh.
  Interventions: Device: Heavy weight Mesh
- Medium weight Mesh (Active Comparator): Intervention: Patients will undergo ventral hernia repair with implantation of a medium weight mesh.
  Interventions: Device: Heavy weight Mesh; Device: Medium weight Mesh

INTERVENTIONS:
Device: Heavy weight Mesh — Patients will undergo ventral hernia repair with heavy weight mesh.
Device: Medium weight Mesh — Patients will undergo ventral hernia repair with medium weight mesh.
  Arms: Medium weight Mesh

SUMMARY:
The purpose of this study is to determine if mesh weight has an impact on postoperative pain, ventral hernia recurrence, incidence of deep wound infection, and overall quality of life following ventral hernia repair with mesh.

DETAILED DESCRIPTION:
Approximately five million laparotomies are performed annually in the United States with upwards of 25% of these patients developing a ventral hernia postoperatively. Despite the prevalence of ventral hernias, the surgical approach to these procedures lacks standardization. In fact, nearly 20%-50% of patients undergoing ventral hernia repair (VHR) will experience a hernia recurrence.

There are several factors that can contribute to ventral hernia recurrence. One of these is the use of prosthetic reinforcement. Although previous studies have shown that the use of mesh during VHR significantly decreases the risk of ventral hernia recurrence, guidelines for the ideal prosthetic material remain unknown. In terms of synthetic mesh, there are proponents that argue the value of medium weight material (40-60 g/m2) in order to combat the risk of postoperative deep surgical site infection and minimize the risk of a "stiff abdomen" or chronic pain syndromes.3-5 On the other hand, however, proponents of a heavier weight material ( > 80 g/m2) argue that its tensile strength leads to a long-term, durable hernia repair with decreased risk of hernia recurrence.

To help determine if mesh weight has an impact on postoperative pain, we propose a registry based, randomized clinical trial (RCT) through the Americas Hernia Society Quality Collaborative (AHSQC). The AHSQC is a multicenter, nationwide quality improvement effort with a mission to improve value in hernia care.6 Data are collected prospectively in the routine care of hernia patients for quality improvement purposes. The information collected in the AHSQC offers a natural repository of information that can be used for research, in addition to its quality improvement purpose. The investigators hypothesize that patients who undergo ventral hernia repair with medium weight mesh will have significantly less pain than those patients who undergo ventral hernia repair using heavy weight mesh one year after operation. Both the intended randomization arms of the study are accepted standard of care practices in use by surgeons.

Specific Aim #1: To determine if the use of a medium weight material leads to a decrease in pain intensity at one year following ventral hernia repair.

Specific Aim #2: To determine if there is a difference in ventral hernia recurrence at one year following surgery.

Specific Aim #3: To determine if there is a difference in the rate of deep surgical site infection at 30-days following surgery between the two mesh types.

Specific Aim #4: To determine if there is a difference in the quality of life between the two groups at one year following surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Will undergo a single-stage, open, retromuscular ventral hernia repair
* CDC Wound Class 1
* Able to achieve midline fascial closure
* Hernia defect width less than or equal to 20 centimeters (measured intraoperatively)
* Able to tolerate general anesthesia
* Able to give informed consent

Exclusion Criteria:

* Patients who are less than 18 years of age
* Patients who undergo emergent ventral hernia repair
* Patients who undergo laparoscopic or robotic ventral hernia repair
* Patients with CDC Wound Class 2, 3, or 4
* Patients who are unable to undergo successful retromuscular mesh placement or who cannot achieve midline fascial closure
* Patients who undergo staged repair of their ventral hernia
* Patients who are unable to give informed consent
* Patients who cannot tolerate general anesthesia
* Patients who are pregnant at the time of surgical intervention

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Rosen, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared, rather the results of the aggregate groups of patients will be shared.

REFERENCES:
- [Derived] Krpata DM, Petro CC, Prabhu AS, Tastaldi L, Zolin S, Fafaj A, Rosenblatt S, Poulose BK, Pierce RA, Warren JA, Carbonell AM, Goldblatt MI, Stewart TG, Olson MA, Rosen MJ. Effect of Hernia Mesh Weights on Postoperative Patient-Related and Clinical Outcomes After Open Ventral Hernia Repair: A Randomized Clinical Trial. JAMA Surg. 2021 Dec 1;156(12):1085-1092. doi: 10.1001/jamasurg.2021.4309. PMID 34524395

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heavy Weight Mesh | Medium Weight Mesh
Started | 173 | 177
Completed | 173 | 177
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Heavy Weight Mesh: Intervention: Patients will undergo ventral hernia repair with implantation of a heavyweight mesh.
  Heavyweight Mesh: Patients will undergo ventral hernia repair with heavweight mesh.
- Medium Weight Mesh: Intervention: Patients will undergo ventral hernia repair with implantation of a mediumweight mesh.
  Heavyweight Mesh: Patients will undergo ventral hernia repair with heavweight mesh.
  Mediumweight Mesh: Patients will undergo ventral hernia repair with mediumweight mesh.
- Total: Total of all reporting groups
Arm/Group | Heavy Weight Mesh | Medium Weight Mesh | Total
Number analyzed (Participants) | 173 | 177 | 350
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.15 (11.35) | 59.31 (11.36) | 59.23 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 91 | 175
  Male | 89 | 86 | 175
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 173 | 177 | 350

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: Pain Scores will be measured using the NIH Promis 3A Pain Scale. PROMIS® Pain Intensity 3A is a three-question instrument developed to measure the range of pain experienced in the week prior to assessment. The raw score (3-15) is converted into a T-score where 50 (SD 10) represents the average of people with at least mild pain, higher numbers (maximum 71.8) represent higher than average pain, and the lowest score (30.7) represents no pain.
Time Frame: One Year Postoperatively
Measure: Median (Inter-Quartile Range); unit: T-Score
Arm/Group | Heavy Weight Mesh | Medium Weight Mesh
Number analyzed (Participants) | 173 | 177
T-Score | 30.7 [30.7 to 43.5] | 30.7 [30.7 to 40.2]

2. Secondary Outcome: Number of Subjects With Hernia Recurrence
Description: Hernia recurrence will be determined using the Ventral Hernia Recurrence Inventory.
Time Frame: One Year Postoperatively
Population: All subjects for both arms were assessed for hernia recurrence, numbers reported below are the number who had recurrence through the following methods of assessment. Some subjects will be in multiple categories
Measure: Number; unit: participants
Arm/Group | Heavy Weight Mesh | Medium Weight Mesh
Number analyzed (Participants) | 173 | 177
participants
  Physical Exam | 2 | 4
  Hernia Recurrence Inventory (HRI)- assessed by subject answering "Yes" to bulge on questionnaire | 52 | 62
  Radiographic- assessed using CT scan | 3 | 3
  Composite Hernia Recurrence (Consensus)- Saying yes to bulge, or having a hernia on imaging or exam | 14 | 13
  Composite Hernia Recurrence (max Sn) includes subjects answering bulge yes and no further follow up | 42 | 48
  Composite Hernia Recurrence (max Sp) includes subjects with only imaging or clinical exam | 3 | 4

3. Secondary Outcome: Deep Wound Infection
Description: The occurrence of a deep wound infection will be determine based on physical examination and/or computed tomography scanning.
Time Frame: 30-Days Postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Heavy Weight Mesh | Medium Weight Mesh
Number analyzed (Participants) | 173 | 177
Participants | 3 | 5

4. Secondary Outcome: Quality of Life Scores
Description: Quality of life will be measured using the HerQLes quality of life questionnaire. HerQLes is a twelve-question instrument developed to evaluate quality of life and function as it pertains to the abdominal wall. It is converted into a 0-100 scale with 0 representing poor abdominal wall function, and 100 excellent function.
Time Frame: One Year Postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Heavy Weight Mesh | Medium Weight Mesh
Number analyzed (Participants) | 173 | 177
score on a scale | 90 [67.92 to 96.67] | 86.67 [65 to 93.33]

ADVERSE EVENTS:
Time Frame: 1 year following surgery for hernia repair
Arm/Group | Heavy Weight Mesh | Medium Weight Mesh
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/177
Serious Adverse Events (participants affected / at risk) | 12/173 | 17/177
Other Adverse Events (participants affected / at risk) | 46/173 | 67/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heavy Weight Mesh (N=173) | Medium Weight Mesh (N=177)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pulmonary Embolism (Vascular disorders) | 2 (2) | 6 (6)
Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Excessive Bleeding (Surgical and medical procedures) | 2 (2) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heavy Weight Mesh (N=173) | Medium Weight Mesh (N=177)
Bleeding (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Bowel Obstruction (Gastrointestinal disorders) | 8 (8) | 4 (4)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Colon Cancer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 18 (18) | 31 (31)
Infection- not otherwise specified (Infections and infestations) | 4 (4) | 9 (9)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 1 (1)
Seroma (General disorders) | 3 (3) | 7 (7)
Surgical Site Infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 4 (4)
Wound Dehiscence (General disorders) | 1 (1) | 4 (4)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT03082391/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03082391/ICF_001.pdf